CLINICAL TRIAL: NCT00372034
Title: The Effect of Punctal Plugs on Tear Volume and Osmolality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRRP2005-018
Record Dates: First submitted 2006-09-03; First posted 2006-09-06 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Dry Eye Syndromes
Keywords: contact lenses; intolerance; punctal plugs; tear volume; Intolerance to contact lens wear due to dryness symptoms
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Device: Temporary Collagen Inserts

SUMMARY:
The purpose of this study is to evaluate the role of tear volume in discomfort and dryness sensations during contact lens wear, and the possible influence on osmolality and ocular surface sensitivity.

DETAILED DESCRIPTION:
50% of contact lens wearers have dryness/discomfort during contact lens wear. Significant decreases in lipid layer and tear film break up time during contact lens wear have been reported, leading to excessive evaporation, reduced tear volume and an increase in osmolality.

Similar tear film changes occur with Dry Eye Disease. A commonly used therapy in treating dry eye is the insertion of punctal plugs to increase tear volume and ease dry eye symptoms. Punctal plugs block the tear drainage system, and often increase tear stability, and improve ocular surface health.

This study will evaluate the role of tear volume in discomfort and dryness sensations during contact lens wear, and the possible influence on osmolality and ocular surface sensitivity. Collagen punctal plugs will be used for this study, as these allow a temporary (3-14 days) occlusion of the ocular drainage system, are easily removed if necessary and are inserted with minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

Exclusion Criteria:

* Corneal refractive surgery
* Contraindications to contact lens wear
* Latex allergy
* Corneal hypoesthesia
* Active corneal infection
* Acute or sub-acute inflammation or infection of the anterior chamber of the eye

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Ocular comfort after 6 hours of contact lens wear
Dryness sensation after 6 hours of contact lens wear
Tear film volume before and after 6 hours of contact lens wear

SECONDARY OUTCOMES:
Objective ocular sensitivity after 6 hours of contact lens wear
Tear film and contact lens osmolality after 6 hours of contact lens wear

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Stahl, Dipl-Optom, Principal Investigator — VisionCRC, School of Optometry and Vision Science, Institute for Eye Research
Locations (1):
- Vision CRC, Institute for Eye Research, School of Optometry and Vision Science, Sydney, New South Wales, Australia